CLINICAL TRIAL: NCT06591065
Title: The Effect of Yoga Education on the Cognitive Status of Performing Arts Students: A Cross-Sectional Study
Brief Title: The Effect of Yoga Education on the Performing Arts Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alanya Alaaddin Keykubat University (Other)
Responsible Party: Principal Investigator, Ayça Araci, PHD, Physiotherapist,PhD, Alanya Alaaddin Keykubat University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 168074
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Yoga; Postural Awareness; Performance Anxiety; Theater; Performing Arts
MeSH Terms: interventions — Control Groups; salicylhydroxamic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral: Yoga Flow (Experimental): The experimental group underwent yoga training conducted by a physiotherapist
  Interventions: Behavioral: Yoga Flow; Other: Controlled
- Controlled Group (No Intervention): The control group did not receive any yoga training

INTERVENTIONS:
Behavioral: Yoga Flow — The study participants were subjected to an intervention comprising hatha yoga sessions conducted twicw weekly over an twelve weeks period, with each session lasting 60 minutes.
  Arms: Behavioral: Yoga Flow
Other: Controlled — The control group did not receive any yoga training
  Other Names: Sham
  Arms: Behavioral: Yoga Flow

SUMMARY:
Objectives. The objective of this study is to examine the effects of yoga exercises on the postural habits and cognitive statutes of the theater students enrolled in the Faculty of Fine Arts, Department of Performing Arts.

Method. A total of 30 volunteers were included in the study, with 15 assigned to the control group and 15 to the experimental group. The efficacy of yoga training was evaluated using pre- and post-intervention scales. The Pittsburgh Sleep Quality Index (PSQI), Postural Habit (P. Habit) and Awareness (P. Awareness) scales, and the Çarkcı Theatre Performance Anxiety Scale (Çr. Theatre Performance Anxiety Scale) were employed for this purpose. Training was conducted twice weekly for a period of 12 weeks.

DETAILED DESCRIPTION:
Yoga is regarded as a mind-body exercise. It emphasizes the interconnection between the body, mind, and spirit and their significance in all facets of personal growth and well-being. It encompasses a diverse array of postures, exercises, breathing techniques, and meditation practices. The fundamental premise underlying these exercises is the notion that an individual's physiological state can influence their emotional, cognitive, and attitudinal processes.

The term "mindfulness" refers to an individual's capacity to engage with their experience in a deliberate manner, with a focus on the present moment. The term "mindfulness" is defined as the act of accepting and approving the present moment without allowing it to be influenced by past experiences or future expectations. The term "active exploration" is used to describe a range of operations, including selection, grasping the foundation, simplification, abstraction, analysis and synthesis, completion, verification, comparison, and problem solving. These processes are not indicative of any specific mental function; rather, they represent the training of cognitive material at any level of the human and animal mind. The prevailing view is that art is a cognitive process and a valuable tool for experimental research, particularly in demonstrating the multiple cognitive abilities that children possess. Body awareness entails the conscious observation of bodily sensations and the cultivation of proprioceptive consciousness. In addition, it is closely related to and strongly linked with the postural awareness structure. The human body is susceptible to a multitude of factors that can influence its posture. These encompass physical, physiological, emotional, and environmental elements. Daily routines and behavioral patterns frequently result in deviations from the optimal body position, leading to alterations in posture. The development of poor posture habits can result in alterations to muscle tone and body alignment, which may subsequently give rise to the formation of poor posture patterns and generalized body asymmetry. It is crucial to be aware of improved ergonomics in order to prevent the onset of musculoskeletal disorders associated with poor posture. An understanding of posture can facilitate the implementation of changes in posture habits.

Performance anxiety is an emotional state that causes a decrease in students' performances due to the fear of being negatively evaluated by instructors in competitive situations, such as exams or concerts, or in situations where their proficiency is tested, such as in musical performances. In this context, the most important factors affecting stage performance can be summarized as motivation, self-determination, difficulty-skill balance, social-physical anxiety concepts. Indeed, for an individual to achieve success on the stage, it is essential to possess a high level of motivation, a distinctive determination, a balanced perception of the level of difficulty and skill required for the role, and a healthy level of social physical anxiety. Sleep quality is a significant factor in cognitive and emotional functioning, and its impairment can have a detrimental impact on an individual's social life and general health status. The study conducted by İyigün et al. underscores the importance of healthy self-determination processes and sleep quality as key determinants of the quality of life of students. People with sleep disorders can gain a healthy sleep cycle by addressing their mental, emotional and physical treatment needs with exercise practices. These exercise practices include strengthening, stretching, Pilates, and yoga exercises. The therapeutic effects of yoga exercises are produced through physiological mechanisms, with significant benefits for physical and emotional health. The practices associated with yoga have been observed to extend to the musculoskeletal system, connective tissues, and mental focus. This results in the acquisition of physical flexibility, which allows the player to utilize the various parts of the body in a more optimal manner. An actor with high body and posture awareness can analyze how to apply the body form desired by the director or role, use it functionally, and be more successful in maintaining continuity.

It is hypothesized that this situation can positively affect the level of anxiety. The exercises that the players perform, particularly those designed to relax them, will prevent the development of unnecessary muscle tension. They will also facilitate increased self-control over their bodies, expand their range of movement on the stage, and provide integrity, precision, comfort, and harmony in movements. It is anticipated that the actor, who has been initiated into the practice of yoga, will demonstrate an understanding of the psychological challenges associated with performance anxiety. Additionally, they will exhibit an awareness of the scene in which they are engaged and a capacity to safeguard their physical well-being through the development of postural awareness, thereby mitigating potential physical and ergonomic risks. The objective of the stage artist is to recreate the reality of life on the stage. In order to achieve this, it is essential that they pay attention to their body, motivation, and musculoskeletal system. However, it is also crucial to consider the physical ergonomic risks that may arise when performing. The field of physical ergonomics is concerned with the physiological responses of the human body to physical work activities, also known as work physiology, as well as the impact of physical dimensions on an employee's abilities, which is referred to as anthropometry. In this instance, it can be posited that the manner in which an individual presents themselves on stage, the style of expression they employ, and their overall demeanor are all influenced by body ergonomics. In contrast to the visual arts, where the majority of ergonomic hazards in the workplace are associated with toxic substances, musculoskeletal issues related to occupational activities have been a significant area of concern for performing artists. In studies of dancers and instrumental musicians, the vast majority of subjects reported both acute and chronic disabling musculoskeletal disorders.

The principal objective of this study was to reveal the effect of yoga exercises on posture habits and awareness, sleep quality and stage performance anxiety in theater students enrolling at the Faculty of Fine Arts, Department of Performing Arts.

ELIGIBILITY:
Inclusion Criteria:

* the ages must be between in 19 and 26.
* Healthy subjects: Indication that participants who do not have a disease or condition.

Exclusion Criteria:

* Cancer
* Hypertension
* Fracture
* Mental disorders
* Risk of pregnancy
* Pregnancy

Ages: 19 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Postural Habit and Awareness Scale | immediately post intervention
  The final iteration of the Postural Habits and Awareness Scale (PHAS) comprises 19 items, which are evaluated on a 5-point Likert scale. Each item on the scale is scored on a Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Seven items are reverse-coded. The maximum score for postural habits is 35, the maximum score for postural awareness is 60, and the maximum possible score is 95. A high score indicates good posture and awareness. Items related to postural habits pertain to expressions regarding the posture that one prefers in activities of daily living, such as standing, sitting, lying down, shopping, and carrying things.
Pittsburgh Sleep Quality Index | immediately post intervention
  The Pittsburgh Sleep Quality Index (PSQI) comprises a total of 24 questions. Of these, 19 are self-assessment questions, while the remaining five are answered by the individual's spouse or roommate.The total score ranges from 0 to 21. A high total score is indicative of poor sleep quality.
Theater Undergraduate Students Performance Anxiety Scale: | immediately post intervention
  The scale was developed to determine the extent of performance anxiety and the level of experience with examinations and performances among undergraduate students enrolled in the Conservatory Theater Department. The Performance Anxiety Scale for Marine Engineering Theater Undergraduate Students consists of 19 items, is five-factor-based, and is designed in a 5-point Likert type. These items, prepared in a 5-point Likert format, are evaluated on a scale ranging from strongly disagree (1 point) to strongly agree (5 points). The lowest score that can be obtained from the scale is 19, indicating a very low level of performance anxiety. The highest score that can be obtained from the scale is 95, indicating a very high level of performance anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Ayça ARACI, Phd, Study Director — Alanya Alaaddin Keykubat University
Locations (1):
- Alanya Alaaddin Keykubat Üniversity, Antalya, Alanya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No